CLINICAL TRIAL: NCT01992211
Title: Randomized, Open, Cross-over, Single Dose Study to Evaluate the PK, Safety/Tolerability of BCWP_C003 Compared to Coadministration of Rosuvastatin and Metformin SR, and the Food Effect on the PK of BCWP_C003 in Healthy Volunteers
Brief Title: Evaluating of Pharmacokinetic Profile of BCWP_C003 and Co-administration of Rosuvastatin and Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BC World Pharm Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: BCWP1202_102
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Metformin

STUDY DESIGN:
Intervention Model Description: 6 x 3
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Treatment Sequence 1(ABC) (Experimental): Participant will be co-administered a single oral dose of Rosuvastatin 10mg and Metformin SR 1000mg under Fed condition on 1Day.
  Participant will be administered a single oral dose of BCWP_C003 under Fasting condition on 8Day.
  Participant will be administered a single oral dose of BCWP_C003 under Fed condition on 15Day.
  Interventions: Drug: Rosuvastatin; Drug: Metformin; Drug: BCWP_C003
- Treatment Sequence 2(ACB) (Experimental): Participant will be co-administered a single oral dose of Rosuvastatin 10mg and Metformin SR 1000mg under Fed condition on 1Day.
  Participant will be administered a single oral dose of BCWP_C003 under Fed condition on 8Day.
  Participant will be administered a single oral dose of BCWP_C003 under Fasting condition on 15Day.
  Interventions: Drug: Rosuvastatin; Drug: Metformin; Drug: BCWP_C003
- Treatment Sequence 3(BAC) (Experimental): Participant will be administered a single oral dose of BCWP_C003 under Fasting condition on 1Day.
  Participant will be co-administered a single oral dose of Rosuvastatin 10mg and Metformin SR 1000mg under Fed condition on 8Day.
  Participant will be administered a single oral dose of BCWP_C003 under Fed condition on 15Day.
  Interventions: Drug: Rosuvastatin; Drug: Metformin; Drug: BCWP_C003
- Treatment Sequence 4(BCA) (Experimental): Participant will be administered a single oral dose of BCWP_C003 under Fasting condition on 1Day.
  Participant will be administered a single oral dose of BCWP_C003 under Fed condition on 8Day.
  Participant will be co-administered a single oral dose of Rosuvastatin 10mg and Metformin SR 1000mg under Fed condition on 15Day.
  Interventions: Drug: Rosuvastatin; Drug: Metformin; Drug: BCWP_C003
- Treatment Sequence 5(CAB) (Experimental): Participant will be administered a single oral dose of BCWP_C003 under Fed condition on 1Day.
  Participant will be co-administered a single oral dose of Rosuvastatin 10mg and Metformin SR 1000mg under Fed condition on 8Day.
  Participant will be administered a single oral dose of BCWP_C003 under Fasting condition on 15Day.
  Interventions: Drug: Rosuvastatin; Drug: Metformin; Drug: BCWP_C003
- Treatment Sequence 6(CBA) (Experimental): Participant will be administered a single oral dose of BCWP_C003 under Fed condition on 1Day.
  Participant will be administered a single oral dose of BCWP_C003 under Fasting condition on 8Day.
  Participant will be co-administered a single oral dose of Rosuvastatin 10mg and Metformin SR 1000mg under Fed condition on 15Day.
  Interventions: Drug: Rosuvastatin; Drug: Metformin; Drug: BCWP_C003

INTERVENTIONS:
Drug: Rosuvastatin — Participants will be co-administered a single oral dose of Rosuvastatin 10mg and Metformin SR 1000mg under Fed condition.
  Other Names: Crestor 10mg(Rosuvastatin)
Drug: Metformin — Participants will be co-administered a single oral dose of Rosuvastatin 10mg and Metformin SR 1000mg under Fed condition.
  Other Names: Glucophage XR 1000mg(Metformin)
Drug: BCWP_C003 — Participant will be administered a single oral dose of BCWP_C003 under Fasting condition or Fed condition according to sequence.
  Other Names: Rosuvastatin and Metformin

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic Profile and Safety/Tolerability of BCWP_C003 compared to Co-Administration of Crestor 10mg and Glucophage XR 1000mg, and to evaluate the food effect of Pharmacokinetic profile of BCWP_C003 after administration.

DETAILED DESCRIPTION:
Clinical Trials to Evaluate the Pharmacokinetic Profiles and Safety/Tolerability of BCWP_C003 Formulation compared to Coadministration of Rosuvastatin and Metformin SR Formulation, and to Evaluate the Effect of Food on the Pharmacokinetic Profile of BCWP_C003 after Single Oral Administration to Healthy Male Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male Volunteer, age 19 to 45 years at the time of screening
* Body weight is not less than 55kg, not more than 90kg and the result of Body Mass Index(BMI) is not less than 18.5, not more than 25.0
* Subject who has no congenital, chronic disease, and no disease symptom or finding in medical examination result
* Subject who comprehended the purpose, contents of the study, property of clinical drug and signed the informed consent to participate in the trial having the willingness

Exclusion Criteria:

* Subject who has history of hypersensitivity reaction for relevant drug(statin, biguanide) or clinically significant hypersensitivity reaction
* Subject who has history or presence of clinically disease in liver, kidney, gastrointestinal tract, respiratory system, musculoskeletal, endocrine system, mental disorder, blood-tumor, cardiovascular. Particulary, subject who has bleeding disorder or tend to be bleeding with bruised easily
* Subject who has family history of hereditary muscular disorder or muscular side effect
* Subject who has history of gastrointestinal tract disorder which can affect the drug absorption or surgery(excluding appendectomy, hernia surgery)
* Subject who had taken diagnosis with peptic ulcer within 2 month prior to the drug administration
* Subject who has results of clinical laboratory test as follows :

  * AST, ALT level exceed the normal range more than 1.5 times
  * Total bilirubin level exceed the normal range more than 1.5 times
  * Creatinine clearance under 60mL/min calculated by MDRD
* In the vital sign, systolic blood pressure is more than 150mmHg, less than 90mmHg or diastolic blood pressure is more than 95mmHg, less than 50mmHg
* Subject who has presence or history of drug abuse, or positive screening for drug abuse

  → Alcohol abuse defines to drink over 21 unit/week(alcohol 1unit = 10g = 12.5 mL) persistingly
* Subject who participated in another clinical trial within 3 month prior to the drug administration
* Subject who had taken medicine(Barbital etc) related drug metabolizing enzyme induction or inhibition within 1 month prior to the drug administration
* Subject who had taken prescription drug or oriental medicine within 2 weeks or OTC drug or vitamin formulation within a week prior to the drug administration
* Subject who had a diet which can affect the absorption, distribution, metabolism or elimination of Rosuvastatin/Metformin (Particulary, Grapefruit - within 48h prior to the drug administration)
* Subject who donated whole blood within 2 month or component blood within 1 month prior to the drug administration
* Subject who smokes more than 10 cigarettes per day
* Subject who has positive HBsAg, HCV Ab or HIV Ab
* Subject who is judged to be ineligible by principal investigator or sub-investigator according to various test results

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Rosuvastatin AUClast | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  Rosuvastatin AUClast
Rosuvastatin Cmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  Rosuvastatin Cmax
Metformin AUClast | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  Metformin AUClast
Metformin Cmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  Metformin Cmax

SECONDARY OUTCOMES:
N-desmethyl rosuvastatin Cmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  N-desmethyl rosuvastatin Cmax
N-desmethyl rosuvastatin AUClast | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  N-desmethyl rosuvastatin AUClast
N-desmethyl rosuvastatin AUCinf | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  N-desmethyl rosuvastatin AUCinf
Rosuvastatin, N-desmethyl rosuvastatin, Metformin AUCinf | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  Rosuvastatin, N-desmethyl rosuvastatin, Metformin AUCinf
Rosuvastatin, N-desmethyl rosuvastatin, Metformin Tmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  Rosuvastatin, N-desmethyl rosuvastatin, Metformin Tmax
Rosuvastatin, N-desmethyl rosuvastatin, Metformin t1/2 | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  Rosuvastatin, N-desmethyl rosuvastatin, Metformin t1/2
Rosuvastatin, N-desmethyl rosuvastatin, Metformin Vz/F | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  Rosuvastatin, N-desmethyl rosuvastatin, Metformin Vz/F
Rosuvastatin, N-desmethyl rosuvastatin, Metformin CL/F | pre-dose, post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36, 48, 72h
  Rosuvastatin, N-desmethyl rosuvastatin, Metformin CL/F

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD. PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No